CLINICAL TRIAL: NCT02460536
Title: Attention Bias Modification Treatment (ABMT) for Anxiety Disorders in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience, Head School of Psychological Sciences, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009341
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Disorders
Keywords: attention bias modification treatment; attention training; anxiety disorders; clinical trials
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Attention Bias Modification treatment (ABMT) (Experimental): Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli using threat and neutral face stimuli.
  Interventions: Behavioral: Attention Bias Modification treatment (ABMT)
- Exposure only +ABMT (Active Comparator): Identical discrimination task including exposure to a single threat or neutral face stimulus in each trial.
  Interventions: Behavioral: Exposure only +ABMT
- Attention training only +ABMT (Active Comparator): Attention training via repeated trials of a dot-probe task using non-emotional stimuli.
  Interventions: Behavioral: Attention training only +ABMT
- Placebo group (Placebo Comparator): Identical discrimination task including a single non-emotional stimulus in each trial.
  Interventions: Behavioral: Placebo group

INTERVENTIONS:
Behavioral: Attention Bias Modification treatment (ABMT) — Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli using threat and neutral face stimuli.
  Arms: Attention Bias Modification treatment (ABMT)
Behavioral: Exposure only +ABMT — Identical discrimination task including exposure to a single threat or neutral face stimulus in each trial.
  Arms: Exposure only +ABMT
Behavioral: Attention training only +ABMT — Attention training via repeated trials of a dot-probe task using non-emotional stimuli.
  Arms: Attention training only +ABMT
Behavioral: Placebo group — Identical discrimination task including a single non-emotional stimulus in each trial.
  Arms: Placebo group

SUMMARY:
Attention biases in threat processing have been assigned a prominent role in the etiology and maintenance of anxiety disorders. Attention Bias Modification Treatment (ABMT) utilizes computer-based protocols to implicitly modify biased attentional patterns in anxious patients. This is a double-blind randomized controlled trial of ABMT for clinically anxious 10-18 year-olds. Participants will be assessed using clinical interviews and parent- and self-rated questionnaires before, in the middle and after twelve sessions of ABMT or control groups, and again at ten-week follow-up. Outcome measures will be anxiety symptoms and depression as measured by gold standard questionnaires as well as structured clinical interviews with youth and their parents. Attentional threat bias, Attentional control and interpretation of ambiguous information will also be measured to explore potential mediators of ABMT's effect on anxiety. The investigators expect the findings to inform pathways to treatments for anxious children and to provide initial information on mechanisms of ABMT efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of GAD, SOP, or SAD.
* Co-morbid attention deficit hyperactivity disorder (ADHD) or depressive disorders must be treated with medication and stable.
* Tics or impulse control problems must be treated with medication, stable and cause minimal or no impairment.

Exclusion Criteria: To be excluded youth must:

* meet diagnostic criteria for Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders, or Mental Retardation.
* show high likelihood of hurting themselves or others.
* have not been living with a primary caregiver who is legally able to give consent for the child's participation.
* be a victim of previously undisclosed abuse requiring investigation or ongoing supervision.
* be involved currently in another psycho-social treatment.
* have a serious vision problem that is not corrected with prescription lenses.
* have a physical disability that interferes with their ability to click a mouse button rapidly and repeatedly.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in anxiety symptoms - the Pediatric Anxiety Rating (PARS) | 4 weeks, 8 weeks, and 18 weeks (follow-up)
  The PARS assesses global anxiety severity across different anxiety disorders in youth.

SECONDARY OUTCOMES:
Change from baseline in anxiety related emotional disorders symptoms - Child/Parent Version (SCARED-C/P) | 4 weeks, 8 weeks, and 18 weeks (follow-up)
  The SCARED is a 41-item self and parent-report instrument designed to assess anxiety in children and adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel